CLINICAL TRIAL: NCT04601155
Title: Transition of Renal Patients Using AlloSure Into Community Kidney Care
Acronym: TRACK
Status: Completed | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00012
Record Dates: First submitted 2020-09-10; First posted 2020-10-23 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — AlloSure Kidney is a blood test that analyzes SNPs selected across all 22 somatic chromosomes to detect DNA released from a patient's kidney allograft, known as donor-derived cell-free DNA (dd-cfDNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- AlloSure Group: Patients will have quarterly AlloSure cfDNA testing (every 3 months) and DSA as part of their post-transplant surveillance for a period of 5 years. For the quarterly AlloSure tests, approximately 20 mL of blood will be obtained in Streck Cell-Free DNA BCT tubes and shipped to CareDx, Inc. (Brisbane, CA) to analyze the presence of donor-derived cell-free DNA.
  Interventions: Device: AlloSure
- Control Group: The control group was never followed with AlloSure as part of their post-transplant follow-up care. Matched control data will originate from UNOS SRTR data.

INTERVENTIONS:
Device: AlloSure — AlloSure is an analytically validated targeted next-generation sequencing (NGS) assay that uses single-nucleotide polymorphisms (SNPs) to measure the fraction of dd-cfDNA in transplant patients without the need for genotyping either the donor or the recipient.8
  Groups: AlloSure Group

SUMMARY:
Patients undergoing kidney transplantation alone (either de-novo or re-transplant) at a participating hospital are routinely surveyed with interval blood tests as part of standard post-operative care through outpatient consultation. These tests include serum creatinine, blood sugar as well as DSA testing at various intervals. The ability to screen patients to better identify those who may be at risk of developing an adverse event using AlloSure cfDNA is likely to be advantageous, with the potential to improve graft survival and outcomes for transplant patients. The addition of AlloSure to the interventional group will be the focus of this study. Patients will have quarterly AlloSure cfDNA testing (every 3 months) and DSA as part of their post-transplant surveillance for a period of 5 years.Participants will attend outpatient visits/follow-up visits as part of their standard care, these will include appointments where they will have blood tests taken as part of post-transplant surveillance. For AlloSure cfDNA and DSA, blood will be taken quarterly.

ELIGIBILITY:
Inclusion Criteria:

* Participants with single kidney transplant (de-novo or re-transplant) who are ≥ 6 months and ≤ 36 months post-transplant. Participants and will need to have a draw in this time period .
* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 12 years or older.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Participant who is pregnant, lactating or planning pregnancy during the trial.
* Significant hepatic impairment (determined by the PI).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months, or inappropriate for diagnostic monitoring through regular blood sampling.
* < 6 months and > 36 months post-transplant
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Multi-organ transplant (e.g., Kidney-Pancreas).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant patients who are having their transplant follow-up care in community nephrology
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Superior allograft survival | 5 years
  Time to allograft loss, defined as composite of: return to dialysis, re-transplant, death due to allograft failure, and death with functioning allograft.

SECONDARY OUTCOMES:
Assessment of kidney function | 5 years
  Relative change in eGFR from baseline in groups monitored using AlloSure compared to matched control group.
Assessment of immunologic status | 5 years
  Proportion of patients with formation of de-novo DSA antibodies in groups monitored using AlloSure compared to matched control group.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Amicis Research Center, Fairfield, California
  - The Medical Research Group - Fresno, Fresno, California
  - Amicis Research Center, Granada Hills, California
  - Amicis Research Center, Mission Hills, California
  - California Institute of Renal Research (Balboa), San Diego, California
  - Starling Physicians, Hartford, Connecticut
  - George Washington/Medical Faculty Associates Inc., Washington D.C., District of Columbia
  - Physician Consultants of Georgia, Macon, Georgia
  - NANI Research, Hinsdale, Illinois
  - NANI Research, Fort Wayne, Indiana
  - Washington University, St Louis, Missouri
  - PRINE Health, Manhasset, New York
  - Chinatown Kidney, New York, New York
  - Nephrology Associates PC, Queens, Queens, New York
  - Sholer Chris MD, Oklahoma City, Oklahoma
  - Utah Kidney Research Institute, South Ogden, Utah
  - Lynchburg Nephrology Physicians, PLLC, Lynchburg, Virginia
  - Mendez Center for Clinical Research, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No